CLINICAL TRIAL: NCT02782390
Title: Efficacy of Hall Technique in Atypical Lesions on Primary Teeth: Randomized Clinical Trial
Brief Title: Efficacy of Hall Technique in Atypical Lesions on Primary Teeth
Acronym: SLM2078
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty Sao Leopoldo Mandic Campinas (Other)
Responsible Party: Principal Investigator, Jose Carlos P Imparato, PhD, Senior Lecturer, Faculty Sao Leopoldo Mandic Campinas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLM3
Record Dates: First submitted 2016-03-10; First posted 2016-05-25 (Estimated); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Dental Caries
Keywords: Stainless dental crown; Composite Resin; Primary teeth
MeSH Terms: conditions — Dental Caries | interventions — Composite Resins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hall Technique (Experimental): single placement of stainless dental crowns on atypical cavities
  Interventions: Other: Dental Restoration with Stainless Crown
- Composite Resin (Active Comparator): single placement of composite resin on atypical cavities
  Interventions: Other: Dental Restoration with Composite Resin

INTERVENTIONS:
Other: Dental Restoration with Stainless Crown — Lesions allocated to this group will be treated with stainless dental crowns according to the Hall Technique protocol (Evans & Innes, 2010).
  Arms: Hall Technique
Other: Dental Restoration with Composite Resin — Surfaces allocated to this group will be treated with composite resin (Z250, 3M ESPE, USA) according to the manufacturer's instructions.
  Initially, local anesthesia and rubber dam adaptation will be performed. Then, 37% phosphoric acid will be applied on the surface for 15 seconds, followed by spray of water/air for at least 15 seconds. Then, the adhesive system (Single Bond, 3M ESPE, USA) will be applied and light cured according to the manufacturer's instructions. Finally, composite resin (Z250, 3M ESPE, USA) will be applied and light cured according to the manufacturer's instructions.
  Arms: Composite Resin

SUMMARY:
Atypical carious cavities could be defined as carious lesions in more than 2 surfaces of the same tooth. Dental practitioners have shown difficulties related to material's maintenance in such type of cavities and therefore, several treatment options have been used. However, most of them have shown a great failure percentage. A randomized clinical trial will be developed with the objective of assessing the Hall technique in comparison with the composite resin incremental technique in 364 primary molars' atypical carious lesions of children between 4 and 9 years old. Initially, two previously calibrated examiners will perform caries diagnosis by means of visual assessment and intraoral examination. Selected teeth will be randomly allocated into two groups. Teeth in the first group will be submitted to prefabricated stainless steel crowns treatment (Hall technique); and the other, to composite resin incremental technique, which will be always placed under rubber dam isolation. Lesions' clinical and radiographic follow-up will be conducted after 6 and 12 months.

Treatment's efficacy will be assessed by means of four main outcomes:

1. Longevity, marginal adaptation, possible modification in patients' vertical dimension, and caries lesion progression;
2. Patient-focused criteria (satisfaction, discomfort and quality of life impact);
3. cost-efficacy; and
4. Treatment-related parents', children' and operators' perception.

Other variables could be further analysed as secondary outcomes, such as techniques performing time among operators, impact of the socio-economic characteristics on restorations' longevity, and restorations' type impact on the antagonist tooth. Comparisons between groups will be addressed using the Kaplan-Meier survival test as well as Long-Rank test. Cox Regression will be used to enable the assessment of other variables' influence in the results. Significance value of 5% will be adopted for all analysis.

ELIGIBILITY:
Inclusion Criteria:

* children must have at least one molar with atypical caries lesion (involving more than two surfaces);
* parents or legal guardians accept and sign the informed consent form.

Exclusion Criteria:

* children with special needs and/or systematic diseases with oral impairment;
* teeth with spontaneous painful symptoms or necrotized and teeth presenting restorations, sealants, developmental enamel defects, pulp exposure or other signs related to endodontic treatment.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 364 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Clinical longevity of restoration | Change from baseline until 6 and 12 months
  The clinical evaluation will be performed by the non-blinded examiners. The examiner will use the criteria proposed by Innes et al. (2007) for both interventions.

SECONDARY OUTCOMES:
Change in patient's vertical dimension | Baseline, 30 days, 6 and 12 months
  The patient's vertical dimension will be measured with a probe (Williams 14, Hu-Friedy Mfg. Co., United Kingdom) according to the protocol described by van der Zee & van Amerongen (2010).
Antagonist's level of intrusion | Baseline, 6 and 12 months
  The crown of the antagonist tooth to the treated tooth will be measured with a calliper and a ruler in cervico-occlusal direction (starting on the concave region of the gingival margin up to the center of the occlusal edge), as proposed by Miraglia et al. (2002) and Magalhaes et al. (2011).
Treatments' cost-efficacy | Through study completion (12 months)
  The costs of each treatment procedure will be calculated and compared with thresholds values for intervention cost-effectiveness by region, determined by World Health Organization (http://www.who.int/choice/costs/CER_levels/en/).
Clinical caries lesion progression | Baseline, 6 and 12 months
  Clinical examination will be performed by a blinded examiner at baseline, 6 months and 12 months after the treatment. These exams will be performed in accordance with Innes et al. (2007).
Impact on children's quality of life (4-5 years old) | Baseline and 6 months
  The oral health related to quality of life will be measured using the validated questionnaire "Early Childhood Oral Health Impact Scale" (ECOHIS) (Tesch et al., 2008) with 4-5 years old children. It will be applied immediately before the procedure and on 6 months follow-up.
Impact on children's quality of life (6-9 years old) | Baseline and 6 months
  The oral health related to quality of life will be measured using the validated questionnaire "Child Perceptions Questionnaire" (CPQ) with 6-9 years old children (Martins et al., 2009). It will be applied immediately before the procedure and on 6 months follow-up.
Children's perceptions about the treatment | Baseline, 6 and 12 months
  Children's perceptions about the treatment performed will be evaluated using the validated questionnaire "Child's and Parent's Questionnaire About Teeth Appearance" (Furtado et al., 2012). This questionnaire will be applied immediately before the procedure and on 6 and 12 months follow-up.
Children's satisfaction with the treatment | Baseline and 6 months
  The patients' satisfaction about the treatment performed will be evaluated using a scale, as performed by Mattos-Silveira et al. (2014). This scale will be applied immediately after the procedure and on 6 months follow-up.
Children self-reported discomfort | Baseline
  The discomfort of each treatment will be evaluated using the facial scale of Wong-Baker (Wong, Baker, 1998). The patient will be asked to choose the face that is more similar to how she/he felt during the treatment.This answer should be given solely by the child, which means no parental or professional interferences.
Marginal adaptation of the stainless steel crowns | Baseline, 6 and 12 months
  This outcome will be evaluated only with the patients randomized to the Hall Technique. The clinician will evaluate the marginal adaptation according to the criteria described by Sharaf & Farsi (2004).
Radiographical caries lesion progression | Baseline, 6 and 12 months
  Radiographical examination will be performed by a blinded examiner at baseline, 6 months and 12 months after the treatment. These exams will be performed in accordance with Innes et al. (2007).
Biofilm retention of the stainless steel crowns | Baseline, 6 and 12 months
  This outcome will be evaluated only with the patients randomized to the Hall Technique. The clinician will evaluate biofilm retention according to the indice proposed by Silness & Loe (1964), adopted to the primary dentition.
Caregivers' perceptions about the treatment | Baseline, 6 and 12 months
  Caregivers' perceptions about the treatment performed will be evaluated using the validated questionnaire "Child's and Parent's Questionnaire About Teeth Appearance" (Furtado et al., 2012). This questionnaire will be applied immediately before the procedure and on 6 and 12 months follow-up.
Clinicians' perceptions about the treatment | Baseline, 6 and 12 months
  Clinicians' perceptions about the treatment performed will be evaluated using the validated questionnaire "Child's and Parent's Questionnaire About Teeth Appearance" (Furtado et al., 2012). This questionnaire will be applied immediately before the procedure and on 6 and 12 months follow-up.
Caregivers' satisfaction with the treatment | Baseline and 6 months
  The caregivers' satisfaction about the treatment performed will be evaluated using a scale, as performed by Mattos-Silveira et al. (2014). This scale will be applied immediately after the procedure and on 6 months follow-up.
Clinicians' satisfaction with the treatment | Baseline and 6 months
  The clinicians' satisfaction about the treatment performed will be evaluated using a scale, as performed by Mattos-Silveira et al. (2014). This scale will be applied immediately after the procedure and on 6 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carlos P Imparato, Professor, Principal Investigator — Faculty Sao Leopoldo Mandic
Locations (1):
- Faculdade Sao Leopoldo Mandic, Campinas, São Paulo, Brazil

REFERENCES:
- [Background] Casagrande L, Dalpian DM, Ardenghi TM, Zanatta FB, Balbinot CE, Garcia-Godoy F, De Araujo FB. Randomized clinical trial of adhesive restorations in primary molars. 18-month results. Am J Dent. 2013 Dec;26(6):351-5. PMID 24640441
- [Background] Evans D, Innes N. The Hall Technique: A minimal intervention, child centred approach to managing the carious primary molar. A Users Manual. University of Dundee, 3. ed., 2010.
- [Background] Innes NP, Ricketts D, Chong LY, Keightley AJ, Lamont T, Santamaria RM. Preformed crowns for decayed primary molar teeth. Cochrane Database Syst Rev. 2015 Dec 31;2015(12):CD005512. doi: 10.1002/14651858.CD005512.pub3. PMID 26718872
- [Background] van der Zee V, van Amerongen WE. Short communication: Influence of preformed metal crowns (Hall technique) on the occlusal vertical dimension in the primary dentition. Eur Arch Paediatr Dent. 2010 Oct;11(5):225-7. doi: 10.1007/BF03262751. PMID 20932395
- [Background] Miraglia SS, Freitas KB, Pinto JHN. Comparative analyze of the mesion-distal (MD) and gengivo-incisal (GI) distances of the upper central incisors with the instrument Trubyte Tooth Indicator. PGRO - Pós-Grad Rev Odontol 5(2):13-17, 2002.
- [Background] Magalhaes JB, Zavanelli AC, Zavanelli RA. Analysis of facial proportion and its relation with dental form, rest and occlusal vertical dimension between institutionalized students. Rev Odontol UNESP 40(5): 215-221, 2011.
- [Background] Tesch FC, Oliveira BH, Leao A. [Semantic equivalence of the Brazilian version of the Early Childhood Oral Health Impact Scale]. Cad Saude Publica. 2008 Aug;24(8):1897-909. doi: 10.1590/s0102-311x2008000800018. Portuguese. PMID 18709230
- [Background] Martins MT, Ferreira FM, Oliveira AC, Paiva SM, Vale MP, Allison PJ, Pordeus IA. Preliminary validation of the Brazilian version of the Child Perceptions Questionnaire 8-10. Eur J Paediatr Dent. 2009 Sep;10(3):135-40. PMID 19761288
- [Background] Furtado GE, Sousa ML, Barbosa TS, Wada RS, Martinez-Mier EA, Almeida ME. [Perceptions of dental fluorosis and evaluation of agreement between parents and children: validation of a questionnaire]. Cad Saude Publica. 2012 Aug;28(8):1493-505. doi: 10.1590/s0102-311x2012000800008. Portuguese. PMID 22892969
- [Background] Mattos-Silveira J, Floriano I, Ferreira FR, Vigano ME, Frizzo MA, Reyes A, Novaes TF, Moriyama CM, Raggio DP, Imparato JC, Mendes FM, Braga MM. New proposal of silver diamine fluoride use in arresting approximal caries: study protocol for a randomized controlled trial. Trials. 2014 Nov 19;15:448. doi: 10.1186/1745-6215-15-448. PMID 25409545
- [Background] Wong DL, Baker CM. Pain in children: comparison of assessment scales. Pediatr Nurs. 1988 Jan-Feb;14(1):9-17. No abstract available. PMID 3344163
- [Background] Sharaf AA, Farsi NM. A clinical and radiographic evaluation of stainless steel crowns for primary molars. J Dent. 2004 Jan;32(1):27-33. doi: 10.1016/s0300-5712(03)00136-2. PMID 14659715
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Derived] Pascareli-Carlos AM, Tedesco TK, Calvo AFB, Floriano I, Gimenez T, Goncalves MDS, Calumby D, Imparato JCP. Survival rate of the Hall technique compared with resin composite restoration in multi-surface cavities in primary teeth: a 1-year randomized clinical trial. J Appl Oral Sci. 2023 Oct 9;31:e20230048. doi: 10.1590/1678-7757-2023-0048. eCollection 2023. PMID 37820181